CLINICAL TRIAL: NCT01147549
Title: An Open-Label, Single-Centre, Phase I Study to Assess the Excretion, Metabolism and Plasma Pharmacokinetics Following a Single Oral Dose of 60 mg [14C]AZD9668 in Healthy Male Volunteers
Brief Title: Single Oral Dose of 60 mg [14C]AZD9668 in Healthy Male Volunteers
Acronym: ADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0520C00016
Record Dates: First submitted 2010-06-11; First posted 2010-06-22 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: ADME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): [C14]AZD9668
  Interventions: Drug: [C14]AZD9668

INTERVENTIONS:
Drug: [C14]AZD9668 — Oral Solution 60 mg Single Dose

SUMMARY:
The purpose of the study is to characterise the absorption, distribution, metabolism and excretion (ADME) of a single oral dose of [14C]AZD9668.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedure
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Exposed to radiation levels above background of >5 mSv in the last year, >10 mSv over the last 5 years or a cumulative total of >1 mSv per year of life
* History or presence of any clinically significant disease or disorder in the opinion of the investigator
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline in the opinion of the investigator

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose recovered in urine and faeces and total balance | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.
Concentration of total radioactivity in blood and plasma | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.
Plasma concentrations of AZD9668 | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.
Metabolite profiling and identification in plasma and excreta | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.
PK of AZD9668 (Cmax, tmax, t½, AUC, CL/F, Vz/F, MRT, fe, Ae, CLR ) | Samples collected prior to treatment, during treatment and follow-up for a maximum of 14 days.

SECONDARY OUTCOMES:
Adverse Events | Adverse events collected prior to treatment and after treatment including follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, Study Director — AstraZeneca R&D, Wilmington; Tim Mant, Professor, Principal Investigator — Quintiles Drug Research Unit, United Kingdom
Locations (1):
- Research Site, London, United Kingdom